CLINICAL TRIAL: NCT05964231
Title: A Double-blind Randomized Controlled Trial Investigating Associations of Microbiota, Serum Total Antioxidant Capacity and Sleep or Psychiatric Symptoms Before and After the Intake of Psychobiotic Lactobacillus Paracasei
Brief Title: The Intervention of Psychobiotics in Patients With Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-I Wu, Senior Attending Psychiatrist, associate professor, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 112-2314-B-195-008-
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Disorders
Keywords: anxiety; microbiota; psychobiotics
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-treated PS23 (Experimental): Lactobacillus paracasei PS23 heat-treated
  Interventions: Dietary Supplement: Heat-treated PS23
- Placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Heat-treated PS23 — Lactobacillus paracasei PS23 heat-treated, 2caps daily use
  Arms: Heat-treated PS23
Dietary Supplement: Placebo — microcrystalline cellulose, 2caps daily use
  Arms: Placebo

SUMMARY:
The investigators designed this double blind randomized controlled study and will recruit 120 patients 20 to 65 years old, with DSM-5 generalized anxiety disorder or unspecified anxiety disorder. After clinical symptoms and psychological evaluation and blood sampling, a semi-structural interview delivered by a psychiatrist will be established to confirm the DSM-5 diagnosis. The participants will be randomly assigned to the Lactobacillus paracasei PS23 psychotropic probiotic or placebo group. Blood and stool samples will be obtained after consent. The samples will be tested for biochemistry, inflammation index, cytokines, intestinal osmotic pressure, or gut permeability, and a Fitbit fitness watch will be given to measure changes in sleep.

DETAILED DESCRIPTION:
This study aimed to recruit 120 subjects that meet the following inclusion criteria after the approval of the IRB. Those agreed to participate and signed the informed consent will be randomly divided into two groups of the Lactobacillus paracasei PS23 psychobiotics capsule and the placebo. Each group aims to recruit 60 people. The power analysis was conducted using effect size for outcomes of improvements in anxiety from previous studies. Based on a power of 80% and assuming a 30% dropout rate and an alpha level of 0.05, a sample of 120 participants (60 per group) will be required. All results will be analyzed using an intent-to-treat analysis based on treatment assignment, regardless of completion or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20~70 years old
2. Patients perceived that they had anxiety-related complaints, or with any type of anxiety disorders of adjustment disorders referred from the Departments of Psychiatry, Neurology, Internal Medicine, and Family Medicine in Mackay Memorial Hospital.
3. Adult GAD-7 ≥ 8 points (to screen for generalized anxiety disorder) or a DSM-5 diagnosis of generalized anxiety disorder (F41.1) or unspecified anxiety disorder (F41.9)
4. Those who are currently under the treatment of selective serotonin reuptake inhibitors (SSRI) will only be included if their SSRI treatment has been stable or has not been changed for 4 weeks.

Exclusion Criteria:

1. Have taken antibiotics or are receiving antibiotic treatment within one month.
2. Have used probiotic products in powder, capsule or tablet form within two weeks (excluding yogurt, Yakult and other related foods).
3. Patients who have undergone hepatobiliary gastrointestinal surgery (except for colorectal polypectomy and appendectomy).
4. Past or current patients with inflammatory bowel disease.
5. Those with a history of cancer.
6. Those who are allergic to lactic acid bacteria products.
7. Patients with severe depression (Patient Health Questionnaire-9 (PHQ-9) ≧ 20 points), or possible neurocognitive impairments (Mini-Mental States Examination (MMSE)<20), or those that had suicidal ideation noted on item 9 from PHQ-9.
8. Patients with chronic psychiatric diseases who are currently taking drugs to treat acute diseases, organic brain diseases, or newly diagnosed or changed drugs within one month.
9. Those who are receiving parenteral nutrition.
10. Those who are evaluated by the principal investigator to be unsuitable to participate in the research.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Changes from the HAM-A compared to placebo. | change from baseline score at 8 weeks
  Hamilton Anxiety Scale(HAM-A) score changes downwards ≥ 20% indicate significant improvement.

SECONDARY OUTCOMES:
Differences in the Generalized Anxiety Disorder 7-item (GAD-7) compared to placebo. | change from baseline score at 8 weeks
  The GAD-7 is a easy to perform initial screening tool for generalized anxiety disorder, When screening for anxiety disorders, a score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder;Using a cut-off of 8 the GAD-7 has a sensitivity of 92% and specificity of 76% for diagnosis generalized anxiety disorder.
Differences in the State and Trait Anxiety Index (STAI) compared to placebo. | change from baseline score at 8 weeks
  The STAI measures levels of anxiety in the current 'state' or from the 'trait'. Good reliability (0.86~0.95) and sensitivity (0.85) were found and the higher the scores, the severe the levels of anxiety.
Differences in Insomnia Severity index (ISI) compared to placebo. | change from baseline score at 8 weeks
  The ISI is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia.
Differences in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) compared to placebo. | change from baseline score at 8 weeks
  The QLESQ-16 is a valid, reliable self-report instrument for assessing quality of life.
Differences in the The Profile of Mood States (POMS) compared to placebo. | change from baseline score at 8 weeks
  The POMS is a psychological rating scale used to assess transient, distinct mood states.
Differences in Visual Analogue Scale-GI (VAS-GI) compared to placebo. | change from baseline score at 8 weeks
  VAS consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
Changes in blood TAC (Total Antioxidant Capacity) before and after consumption of probiotics | change from baseline score at 8 weeks
  TAC is the biomarker for Oxidative stress.
Changes in blood DHEA-S (Dehydroepiandrosterone sulfate) compared to placebo. | change from baseline score at 8 weeks
  DHEA-S is the biomarker for anti-aging，among the neuroactive steroids, dehydroepiandrosterone (3b-hydroxyandrost-5-ene-17-one, [DHEA]) and its sulfated metabolite DHEA sulfate (DHEAS) have been shown to be potent modulators of neural function, including neurogenesis, neuronal growth and differentiation, and neuroprotection. Highlighting the potential health significance of DHEA and DHEAS in humans, serum concentrations decrease steadily with age, with lowest concentrations present at the time many diseases of aging and neurodegeneration become apparent.
Changes in blood Cortisol compared to placebo. | change from baseline score at 8 weeks
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help: body respond to stress or danger increase your body's metabolism of glucose control your blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by your body to ensure the balance is correct.
Changes in blood High sensitivity CRP (hs CRP) compared to placebo. | change from baseline score at 8 weeks
  High-sensitivity C-reactive protein (hsCRP) is a marker of inflammation that predicts incident myocardial infarction, stroke, peripheral arterial disease, and sudden cardiac death among healthy individuals with no history of cardiovascular disease, and recurrent events and death in patients with acute or stable coronary syndromes.
Improvements and differences compared to placebo on oxidative, inflammation, and stress biomarkers. | change from baseline score at 8 weeks
  Analyses on inflammatory and anxiety measures cytokines including IL-2, IL-6, IL-10, IL-1beta, TNF-alpha, and BDNF will be performed by ELISA tool following the suppliers' protocol (eBioscience, Boston, MA).
Changes zonulin and calprotectin in fecal sample compared to placebo. | change from baseline score at 8 weeks
  The composition of the gut microbiome from stool sample will be examined by Illumina MiSeq Platform. Fecal sample will be washed and prepared with sterile PBS. All samples will be prepared according to the manufacturer's guidelines. Fecal DNA on the V3-V4 regions will be amplified by16s amplicon PCR primers. An online bioinformatics database will be used for the identifications of bacteria and quality filtering.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-I Wu, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan